CLINICAL TRIAL: NCT00594841
Title: A Multicenter Randomized Clinical Trial of Non-operative Versus Operative Treatment of Acute Acromioclavicular Joint Dislocation
Brief Title: Non-operative Versus Operative Treatment of Acute Acromioclavicular Joint Dislocation
Acronym: ACJoint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Orthopaedic Trauma Association (Other); Osteosynthesis & Trauma Care (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC 02-Nov-07; MMES 2008
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Shoulder Dislocation
Keywords: Acromioclavicular Joint; Shoulder dislocation; AC dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Conservative (nonoperative) management of the AC joint dislocation.
  Interventions: Other: Non operative treatment of AC joint dislocation (sling)
- 2 (Experimental): Operative fixation (i.e., ORIF) of the dislocation with a hook plate and screws.
  Interventions: Procedure: Open Reduction Internal Fixation of AC joint dislocation

INTERVENTIONS:
Procedure: Open Reduction Internal Fixation of AC joint dislocation — Definitive surgical treatment (i.e., ORIF) will be performed within 28 days of the injury. In all cases the procedure will be performed by an orthopedic staff surgeon with the assistance of a fellow/resident(s). The operating surgeon will determine the positioning of the patient for surgery. ORIF of the AC joint dislocation will be carried out as follows:
  * Anatomic reduction of the AC joint
  * Definitive fixation with a hook plate and screws
  Arms: 2
Other: Non operative treatment of AC joint dislocation (sling) — Standard protocol for conservative treatment will consist of the implementation of a sling, for shoulder support and patient comfort, for four weeks followed by physiotherapy. Pendulum exercises may be implemented at any time as dictated by the attending surgeon.
  Arms: 1

SUMMARY:
The purpose of this study is to compare non-operative treatment versus operative treatment in patients who suffer a complete, acute acromioclavicular (AC) joint dislocation. This study will show if one method is superior to the other and will also show advantages and disadvantages associated with each treatment method.

DETAILED DESCRIPTION:
All patients presenting to the hospital with a Type III, IV or V acute acromioclavicular (AC) joint dislocation and meeting the eligibility criteria will be approached and asked to enter this prospective, randomized clinical trial. After obtaining consent, the subject will be managed in accordance with one of the two randomized treatment strategies. The first treatment strategy will involve conservative (nonoperative) management of the AC joint dislocation. The second treatment strategy will involve operative fixation (i.e. ORIF) of the dislocation with a hook plate and screws.

The subjects in both treatment groups will receive post-operative care according to the same standards and protocol. The surgeon and research staff will be responsible for study follow-up (clinical and radiological assessment) of the patient on admission (baseline), on discharge from the hospital and at post-operative intervals of six weeks, three months, six months, one year and two years. Primary and secondary outcomes will be monitored at these post-operative intervals.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 16 to 65 years of age
* Grade III (3), IV (4) or V (5) dislocation of the acromioclavicular (AC) joint (evidenced by no contact between the distal clavicle and the acromion as seen in standardized radiographs)
* Closed injury
* AC joint dislocations within 28 days post injury
* Provision of informed consent

Exclusion Criteria:

* Grade I(1), II (2), or VI (6) subluxation/dislocation of the AC joint
* Open AC joint separation
* Scapulothoracic dissociation
* Presence of vascular injury
* Dislocations over 28 days post-injury
* Limited life expectancy due to significant medical co-morbidity
* Medical contraindication to surgery (including pregnancy)
* Inability to comply with rehabilitation or form completion
* Inability to provide informed consent
* Likely problems, in the judgement of the investigators, with maintaining follow-up (i.e., patients with no fixed address, patients not mentally competent to give consent, etc.)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be a patient-oriented, limb-specific, functional measurement questionnaire score (Disabilities of the Arm, Shoulder and Hand - DASH). | 2 years
  2 years for recruitment plus 2 years for follow-up. Total study duration = 4 years

SECONDARY OUTCOMES:
Secondary measures will include radiographic (anatomical reduction and arthritic changes 20) and clinical assessment outcomes. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael D McKee, MD, FRCSC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Canadian Orthopaedic Trauma Society. Multicenter Randomized Clinical Trial of Nonoperative Versus Operative Treatment of Acute Acromio-Clavicular Joint Dislocation. J Orthop Trauma. 2015 Nov;29(11):479-87. doi: 10.1097/BOT.0000000000000437. PMID 26489055